CLINICAL TRIAL: NCT02883244
Title: Effect of Curved Design Soft-Picks on Plaque Accumulation on Patients With Signs of Gingivitis
Brief Title: Curved Soft-Picks on Plaque Accumulation on Patients With Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLP-2015-11-16-1
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2017-05

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Soft-Picks Advanced (Experimental): Device: Curved Soft-Picks
  Interventions: Device: Soft-Picks Advanced
- Floss (Active Comparator): Device: Waxed tape floss
  Interventions: Device: Floss

INTERVENTIONS:
Device: Soft-Picks Advanced — Soft-picks Advanced will be used once a day to clean interdental sites at home.
  Arms: Soft-Picks Advanced
Device: Floss — Floss will be used once a day to clean interdental sites at home.
  Arms: Floss

SUMMARY:
The aim of this study is to evaluate the efficacy of a new interdental cleaning device (Soft-Picks Advanced), as compared to a leading brand floss; and, how ease of use can promote the establishment of a hygienic routine of cleaning interproximal spaces.

DETAILED DESCRIPTION:
The Soft-Picks Advanced has a new curved design allowing a user to easily access to difficult interdental sites, such as spaces between premolars and molars. This study is a single center with parallel design, single blinded, which will randomize eligible subjects into two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and physically able to carry out all study procedures and be available at all times required for participation
* Be able to fully understand and comply with the written and verbal instructions provided
* Provide written Informed Consent
* Be age 18 - 70 years
* Agree to return study materials at the required visit(s)
* Have a minimum of 20 'scorable' teeth (excluding 3rd molars)
* Have more than or equal 10% and less than or equal to 50% Bleeding on Probing (BOP) sites
* Have all Pocket Depth (PD) less than or equal to 4mm
* Have at least 12 qualifying, interproximal sites (6 per side) with closed contacts, without crown or restorations. (See section 5.1.1 'Teeth Selection')
* Be a regular manual toothbrush user for at least 2 months.
* Be a non-smoker for at least 2 years.
* Be willing to abstain from use of chewing gum and consumption of apples, carrots or other hard crunchy foods or thick skinned fruits for 3-6 hours before each visit.
* Be willing to comply with 12-18 hours of no oral hygiene practices

Exclusion Criteria:

* Medical or Dental condition that would be unduly affected by participation in this study, per Investigator Discretion
* Pregnant or nursing, per urine based pregnancy test
* A medical condition requiring antibiotic pre-medication prior to dental appointments
* Diagnosis of Xerostomia
* Any oral or extra oral piercing that interferes with the ability to perform study procedures and/or clinical assessments in the mouth
* Currently undergoing or requiring dental/periodontal treatment, or having had periodontal treatment in the six months preceding the study, where the subject's study participation could present an undue safety risk or obscure the evaluation of study endpoints, per Investigator /Examiner discretion
* Oral surgery within the last 2 months
* A known allergy or sensitivity to products planned for use in this study
* Unwillingness to abstain from all other oral hygiene products other than those prescribed for the duration of the study
* Participation in an oral care study within the previous 90 days
* Are a dental student or dental professional
* Uncontrolled Diabetes
* Current use of antibiotic medications or use within 4 weeks of enrollment
* Presence of heavy deposits of calculus, either supragingival and/or subgingival, per Investigator/Examiner discretion
* Extensive crown or bridge work, rampant decay or excessive gingival recession, per Investigator/Examiner discretion
* Presence of orthodontic bands interfering with efficacy outcome(s) per Investigator/Examiner discretion
* Current use of professionally dispensed bleaching products or use within one month of screening.
* Be an employee, spouse or a relative of an employee of the clinical research site, or a dental products manufacturing, research or marketing firm.
* Chronic treatment with any medication known to affect periodontal status within one month of the screening examination (daily use of 81 mg Aspirin is not exclusionary)
* Have any tooth sites with: > 5mm PD or attachment loss > 3mm, excluding 3rd molars

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Moretti, DDS, MS, Principal Investigator — Clinical Associate Professor and Graduate Program Director
Locations (1):
- Department of Periodontology UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled subjects with signs and symptoms of gingivitis and no or little experience with inter-proximal cleaning device in the single center.
Pre-assignment Details: All subjects received professional prophylaxis and assigned manual toothbrush and dentifrice. Group was assigned 3 weeks or more after professional prophylaxis.
Period: Overall Study
Arm/Group | Floss | Soft-Picks Advanced
Started | 24 | 26
Completed | 24 | 25
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Soft-Picks Advanced | Floss | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (6.9) | 26.9 (8.5) | 26.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 2 | 2
  African American, Asian, Caucasian | 1 | 0 | 1
  American Indian/Caucasian | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Caucasian | 21 | 16 | 37
  Other | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Interproximal Plaque by Modification of the Quigley-Hein Plaque Index at 14 Days
Description: Plaque scores shall be visually assessed at the four (2) tooth surfaces that make up each of the 12 (6 per side) qualifying interproximal test units: mesiobuccal and distobuccal (scale of 0-5, 0 =No debris or stain present on the clinical crown; 5=Plaque coverage over more than two third of the tooth surface). Change = (14 days Score - Baseline Score)
Time Frame: Baseline and 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Soft-Picks Advanced | Floss
Number analyzed (Participants) | 26 | 24
score on a scale | 0.03 (1.02) | -0.07 (1.12)

2. Primary Outcome: Change in Interproximal Plaque by Modification of the Quigley-Hein Plaque Index at 28 Days
Description: Plaque scores shall be visually assessed at the four (2) tooth surfaces that make up each of the 12 (6 per side) qualifying interproximal test units: mesiobuccal and distobuccal (scale of 0-5, 0 =No debris or stain present on the clinical crown; 5=Plaque coverage over more than two third of the tooth surface) Change = (28 days Score - Baseline Score)
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Soft-Picks Advanced | Floss
Number analyzed (Participants) | 25 | 24
score on a scale | 0.04 (1.19) | 0.23 (0.93)

3. Secondary Outcome: Performance (Easy to Use) of an Assigned Product
Description: Subjects record product performance and experience on a diary. Scale of Easy to Use was scored from 1 to 5 (1= Not easy; 5= Very easy).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Soft-Picks Advanced | Floss
Number analyzed (Participants) | 25 | 24
score on a scale | 3.8 (0.21) | 3.37 (0.17)

4. Secondary Outcome: Change in Gingivitis by UNC Modified Gingival Index at 28 Days
Description: Gingiva shall be assessed at 6 sites per tooth: distobuccal, direct buccal, mesiobuccal, distolingual, direct lingual and mesiolingual surfaces (Scale is 0-3: 0 =Normal gingiva (pink, firm, stippled), 3 =Severe inflammation: marked redness and edema, ulceration, tendency to spontaneous bleeding). Change = (28 days Score - Baseline Score)
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Soft-Picks Advanced | Floss
Number analyzed (Participants) | 25 | 24
units on a scale | -0.02 (0.35) | 0.03 (0.37)

5. Secondary Outcome: Change in Gingivitis by Bleeding on Probing at 28 Days
Description: Presence or absence of bleeding within 10 seconds after probing shall be scored at 6 sites per tooth: distobuccal, distal, mesiobuccal, and distolingual, lingual and mesiolingual surfaces. The number of sites where bleeding is recorded is divided by the total number of available sites and multiplied by 100 to express the bleeding on probing as a percentage. Change = (28 days percentage - Baseline percentage)
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: percentage of Bleeding on Probing
Arm/Group | Soft-Picks Advanced | Floss
Number analyzed (Participants) | 25 | 24
percentage of Bleeding on Probing | 7 (21.2) | 13 (17.7)

6. Secondary Outcome: Change in Gingivitis by Probing Pocket Depth at 28 Days
Description: 6 sites per tooth: distobuccal, distal, mesiobuccal, and distolingual, lingual and mesiolingual surfaces: (mm) Change = (28 days measurement - Baseline measurement)
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Soft-Picks Advanced | Floss
Number analyzed (Participants) | 25 | 24
mm | -0.16 (0.21) | 0 (0.23)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Soft-Picks Advanced | Floss
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 1/26 | 5/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soft-Picks Advanced (N=26) | Floss (N=24)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Ingrown toenail (Infections and infestations) | 0 (0) | 1 (1)
Finger dislocating (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Torn hamstring (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. PI shall delay publications for up to 60 days to allow sufficient time to resolve any questions or seek patent protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02883244/Prot_SAP_000.pdf